CLINICAL TRIAL: NCT03359018
Title: Apatinib Mesylate Plus Anti-PD1 Therapy (SHR-1210) in Locally Advanced, Unresectable or Metastatic Osteosarcoma(APFAO)Refractory to Chemotherapy : a Single Institution, Open-label, Phase 2 Trial
Brief Title: Apatinib Plus Anti-PD1 Therapy for Advanced Osteosarcoma
Acronym: APFAO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PKUPH-sarcoma 02
Record Dates: First submitted 2017-11-27; First posted 2017-12-02 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Progression-free Survival; Overall Survival; Clinical Benefit Rate; Toxicity
Keywords: osteosarcoma; advanced; apatinib; PD-1
MeSH Terms: conditions — Osteosarcoma | interventions — apatinib; camrelizumab

STUDY DESIGN:
Intervention Model Description: Every patients will received apatinib 500mg or 250mg orally daily and SHR-1210 3mg/kg (no more than 200mg) iv every 2 weeks until disease progression or intolerance to side effects
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- apatinib plus anti-PD1 therapy arm (Experimental): Every patients will received apatinib 250mg or 500mg orally daily and SHR-1210 3mg/kg (no more than 200mg) iv every 2 weeks until disease progression or intolerance to side effects.
  Interventions: Drug: Apatinib; Drug: SHR-1210

INTERVENTIONS:
Drug: Apatinib — Every patients will received apatinib 250mg or 500mg orally daily according to their body surface area (BSA) until disease progression or intolerance to side effects.
Drug: SHR-1210 — Every patients will received SHR-1210 3mg/kg (no more than 200mg) iv every 2 weeks until disease progression or intolerance to side effects.

SUMMARY:
After standard multimodal therapy, the prognosis of relapsed and unresectable high-grade osteosarcoma is dismal and unchanged over the last decades. We have already finished a prospective trial about apatinib for advanced osteosarcoma(NCT02711007) and find it has a objective response rate of aproximately 45% with median progression-free survival around 5 months. Thus, the investigators explored apatinib activity together with anti-PD1 therapy in order to induce durable response in patients with relapsed and unresectable osteosarcoma after the failure of first-line or second-line chemotherapy.

Apatinib is a small-molecule vascular endothelial growth factors receptor (VEGFR) tyrosine kinase inhibitor, similar to pazopanib, but with a binding affinity 10 times to VEGFR-2 comparing with pazopanib or sorafenib.

SHR-1210 is a humanized anti-PD-1 monoclonal antibody.

DETAILED DESCRIPTION:
Patients more than 11 years with body surface area more than 1.2m2, progressing after standard treatment, will be eligible to receive 250 or 500 mg of apatinib once daily together with SHR-1210 3mg/kg (no more than 200mg) iv every 2 weeks until progression or unacceptable toxicity. The primary end point was progression-free survival (PFS) at 4 months and overall survival(OS). Secondary objectives were clinical benefit rate (CBR), defined as no progression at 6 months and safety.

ELIGIBILITY:
Inclusion Criteria:

* age more than or equal to 11 years;
* diagnosis confirmed histologically and reviewed centrally;
* prior treatment (completed >4 weeks before trial entry) consisted of standard high-grade osteosarcoma chemotherapy agents including doxorubicin, cisplatin, high- dose methotrexate, and ifosfamide; metastatic relapsed and unresectable progressive disease (PD);
* having measurable lesion according to RECIST 1.1;
* Eastern Cooperative Oncology Group performance status 0-1 with a life expectancy >3 months;
* Patients must have adequate organ function (without blood transfusion, without growth factor or blood components support within 14 days before enrollment)as determined by: Hemoglobin ≥ 9 g/dL; Absolute neutrophil count (ANC) ≥1.5×109/L; Platelet count ≥ 75×109/L (for patients with advanced hepatocellular carcinoma), Platelet count ≥ 100×109/L (for patients with advanced gastric cancer); serum albumin ≥2.8 g/dL; serum total bilirubin (TBIL)≤1.5 times the upper limit of normal (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×upper limit of normal(ULN), for subjects with liver metastases, ALT and AST≤5×ULN; Calculated creatinine clearance (CrCl) > 50 mL/min (Cockcroft-Gault formula will be used to calculate CrCl).
* normal or controlled blood pressure;
* Females of childbearing potential (FOCBP), who are not surgically sterile or postmenopausal, must conduct pregnancy test (serum or urine) within 7 days before enrollment, and must not be pregnant or breast-feeding women.
* surgery and/or radiotherapy completion at least 1 month before enrollment.
* Joining the study voluntarily with good compliance.

Exclusion Criteria:

* Patients must not have had prior treatment with camrelizumab or any other PD-L1 or PD-1 antagonists.
* Patients with any active autoimmune disease or history of autoimmune disease, including but not limited to the following: hepatitis, pneumonitis, uveitis, colitis (inflammatory bowel disease), hypophysitis, vasculitis, nephritis, hyperthyroidism, and hypothyroidism, except for subjects with vitiligo or resolved childhood asthma/atopy. Asthma that requires intermittent use of bronchodilators or other medical intervention should also be excluded.
* Concurrent medical condition requiring the use of immunosuppressive medications, or immunosuppressive doses of systemic or absorbable topical corticosteroids. Doses > 10 mg/day prednisone or equivalent are prohibited within 2 weeks before study drug administration. Note: corticosteroids used for the purpose of IV contrast allergy prophylaxis are allowed.
* Known history of hypersensitivity to any components of the camrelizumab formulation, or other antibody formulation.
* Active central nervous system (CNS) metastases with clinical symptoms (including cerebral edema, steroid requirement, or progressive disease). Subjects with brain or meningeal metastases that were previously treated must be clinically stable (magnetic resonance imaging [MRI] at least 4 weeks apart do not show evidence of new or enlarging metastases) and have discontinued immunosuppressive doses of systemic steroids (> 10 mg/day prednisone or equivalent) for at least 2 weeks before study drug administration.
* Patients with other malignant tumor (except cured skin basal cell carcinoma and cervical carcinoma).
* Clinically significant cardiovascular and cerebrovascular diseases, including but not limited to severe acute myocardial infarction within 6 months before enrollment, unstable or severe angina, or coronary artery bypass surgery, Congestive heart failure (New York heart association (NYHA) class > 2), ventricular arrhythmia which need medical intervention, left ventricular ejection fraction(LVEF) < 50%.
* Hypertension and unable to be controlled within normal level following treatment of anti-hypertension agents(within 3 months): systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg.
* Coagulation abnormalities (PT>16s、APTT>43s、TT>21s、Fbg<2g/L), with bleeding tendency or are receiving thrombolytic or anticoagulant therapy.
* Active infection or an unexplained fever > 38.5°C during screening visits or on the first scheduled day of dosing (at the discretion of the investigator, subjects with tumor fever may be enrolled).
* Previous experience abdomen fistula, gastrointestinal perforation, or abdominal abscess within 4weeks.
* Objective evidence of previous or current pulmonary fibrosis history, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonia, pulmonary function damaged seriously etc.
* History of immunodeficiency including seropositivity for human immunodeficiency virus (HIV), or other acquired or congenital immune-deficient disease, or active hepatitis (transaminase does not meet the inclusion, hepatitis B virus (HBV) DNA ≥10⁴ /ml or hepatitis C virus (HCV) RNA≥103 /ml or higher); Chronic hepatitis B virus carriers who HBV DNA<2000 IU/ml(<104/ml), must receive anti-viral treatment throughout the study.
* Any other medical, psychiatric, or social condition deemed by the investigator to be likely to interfere with a subject's rights, safety, welfare, or ability to sign informed consent, cooperate, and participate in the study or would interfere with the interpretation of the results.

Min Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-10-22 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
progression-free survival | up to approximately 24months
  Progression-free survival is defined as time from enrollment to the first occurrence of progression of disease or death from any cause within 63 days of last response assessment.
clinical benefit rate | up to approximately 24months
  clinical benefit rate is defined as the proportion of patients who achieve disease control (objective response and stable disease according to RECIST 1.1).

SECONDARY OUTCOMES:
overall survival | up to approximately 5 years
  overall survival is defined as the duration from date of enrollment to the date of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Guo, M.D.and Ph.D., Principal Investigator — Musculoskeletal Tumor Center of Peking University People's Hospital
Locations (2):
- China (2):
  - Musculoskeletal Tumor Center of Peking University People's Hospital, Beijing
  - Peking University Shougang Hospital, Beijing

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: from completion of the study to study publication

REFERENCES:
- [Background] Xie L, Xu J, Sun X, Tang X, Yan T, Yang R, Guo W. Apatinib for Advanced Osteosarcoma after Failure of Standard Multimodal Therapy: An Open Label Phase II Clinical Trial. Oncologist. 2019 Jul;24(7):e542-e550. doi: 10.1634/theoncologist.2018-0542. Epub 2018 Dec 17. PMID 30559126
- [Background] Xie L, Xu J, Sun X, Tang X, Yan T, Yang R, Guo W. Anorexia, Hypertension, Pneumothorax, and Hypothyroidism: Potential Signs of Improved Clinical Outcome Following Apatinib in Advanced Osteosarcoma. Cancer Manag Res. 2020 Jan 7;12:91-102. doi: 10.2147/CMAR.S232823. eCollection 2020. PMID 32021426
- [Result] Xie L, Xu J, Sun X, Guo W, Gu J, Liu K, Zheng B, Ren T, Huang Y, Tang X, Yan T, Yang R, Sun K, Shen D, Li Y. Apatinib plus camrelizumab (anti-PD1 therapy, SHR-1210) for advanced osteosarcoma (APFAO) progressing after chemotherapy: a single-arm, open-label, phase 2 trial. J Immunother Cancer. 2020 May;8(1):e000798. doi: 10.1136/jitc-2020-000798. PMID 32376724

DOCUMENTS (1):
  • Study Protocol (2017-12-02): https://cdn.clinicaltrials.gov/large-docs/18/NCT03359018/Prot_001.pdf